CLINICAL TRIAL: NCT07354204
Title: Tart Cherries - The Influence on Acute Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: Iprona Lana SpA (Unknown)
Responsible Party: Principal Investigator, Glyn Howatson, Professor Glyn Howatson, Northumbria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 51533
Record Dates: First submitted 2025-09-27; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Recovery
Keywords: Repeated bout effect; exercise recovery; tart cherry; muscle damage

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vistula Tart Cherry (Active Comparator): Supplemented with tart cherries.
  Interventions: Dietary Supplement: Tart Cherry
- Placebo (Placebo Comparator): Supplemented with a calorie matched placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Tart Cherry — 7 day supplementation
  Arms: Vistula Tart Cherry
Other: Placebo — 7 day supplementation
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to compare recovery and impact on acute adaptation conferred by the RBE following eccentric exercise in healthy, active participants.

The main questions it aimed to answer were whether 7 day supplementation with Vistula tart cherries attenuated:

* muscle function
* inflammation
* soreness

Participants will either consume a spray-dried tart cherry supplement or a calorie-matched placebo-control for 7 days, and complete two bouts of eccentric exercise to the elbow flexors. Participants will perform functional tests, be assessed for their perceptual recovery and markers of inflammation and muscle damage via:

* maximal voluntary contractions
* visual analog scales to assess soreness
* blood samples

DETAILED DESCRIPTION:
Participants Twenty-one recreationally active participants (2 females) were recruited for this study; the mean ± SD age, stature and mass were 27 ± 7 years old, 179.5 ± 8.6 cm and 80.86 ± 11.29 kg, respectively. Participants were healthy, non-smoking, with no history of cardiovascular, gastrointestinal, thyroid or renal disease and free from musculoskeletal injuries. Further exclusion criteria stipulated the participants were not to be highly trained or partaking in structured resistance training. Health and training status were determined by a screening questionnaire. Highly trained was defined as completing structured and periodized training and developing towards (within 20%) of maximal or nearly maximal norms within their given sport. Participants were asked to refrain from all exercise five days prior to, and for the duration of testing. The participants were also asked to maintain their habitual diet and to complete a food log to ascertain polyphenols intake, such as fruits & vegetables, fruit juices, nuts and seeds, chocolate and coffee/tea. Further, participants were asked to refrain from non-steroidal anti-inflammatory drugs and nutritional supplements, such as ibuprofen, paracetamol, protein, vitamin C and E. This study received ethical approval from Northumbria University Ethics Committee (reference number: 51533 ).

Experimental Design The study was a double-blind, randomised, placebo-controlled design. Participants were subject to block randomisation to one of two groups to consume either the VTC supplement or a placebo, matched for calorific content. Participants were required to come to the lab on a total of nine occasions, which included a familiarisation (visit 1). Bout 1 (visit 2) and Bout 2 (visit 6) were separated by two weeks. Each damaging bout was followed by 3 consecutive days to record dependent measures, which took place at the same time of day (±2h). The loading phase for the supplement ingestion commenced 4 days prior to the first exercise bout, and continued on the day of the exercise, and for 3 days following the exercise bout. No supplement was consumed before or during bout 2 for either group. Lastly, participants were required to fill in a food diary in the 24 h prior to the damaging bout to monitor food and drink intake and enable replication for subsequent sessions.

Damage Protocol An isokinetic dynamometer (Biodex System 4, New York, NY, USA) was set up as recommended by the manufacturer to test the dominant elbow flexors. The participant's position was stabilised using a pelvic strap and two shoulder straps to minimise mechanical assistance from other body parts. The final position of the dynamometer seat and power head were recorded and replicated for each participant's to ensure consistency on subsequent days. Joint position and range of motion was monitored throughout by extracting data from the dynamometer to an analogue-to-digital converter (Micro 1401, Cambridge Electronic Design; CED, Cambridge, UK) to ensure on return visits each participant was placed in an identical position (recorded on Spike2, v7.12; CED, Cambridge, UK). In accordance with previous recommendations [50], dynamometer readings were corrected for the gravity acting upon limb mass. The dynamometer was set to an angular velocity of 30 degrees/s-1 in the passive mode and participants were instructed to resist maximally from full elbow flexion through the whole range of motion until full extension was achieved. Each participant completed 40 (five sets of eight repetitions; each set separated by 90 s rest) maximal lengthening contractions of the elbow flexors. Previous research utilising a protocol of the same intensity but varying in volume-both lower and higher-has successfully induced muscle damage. Visual feedback from the dynamometer and standardised strong verbal encouragement from the investigator was given during the damaging exercise to encourage maximal effort. This was performed on visit 2 (bout 1) and visit 6 (bout 2) of the study.

Supplementation The participants consumed either a placebo or a TC spray-dried extract made from the Vistula cultivar (Iprona Lana SpA, South Tyrol, Italy), in the form of capsules, twice per day for a period of eight days. The supplementation period was selected to replicate similar the loading phases of TC supplementation reported in previous work. The dose increased on the day of the damaging bout 1. The rationale for the dose increase was based on previous research that showed increased bioavailability of circulating anthocyanin and polyphenols, which were considered important in the current study to reduce the additional negative effects associated with EIMD. The participants were required to consume a lower dose (73.5 mg of anthocyanins) for the first four days, then consume a higher dose (132.3 mg of anthocyanins) for the remaining four days (day of damage protocol, 24, 48 and 72 h post). The loading dose was determined by replicating similar volumes of reported anthocyanin content from previous studies that used powdered TC supplement. The higher dose was doubled, similarly to research which have observed differences in dose-response relationship studies. No supplement was consumed before or during bout 2 to ascertain the influence of VTC on the adaptive response expected following Bout 2.

Functional Performance and Perceptual Variables Dependent variables were recorded at baseline, 24-, 48- and 72-h post the damage protocol (for both Bout 1 and 2), measures of functional performance and perceptual variables were used to assess the fatigue and recovery after an isolated muscle damage protocol.

Maximal Voluntary Contraction Participants performed a warm-up on the aforementioned dynamometer, which consisted of three submaximal contractions at a participant perceived intensity of 30, 50 and 70% MVC. MVC was determined at a joint angle of 45° of flexion from full extension, following an identical method previously reported from our laboratory (CV < 5%). Three isometric contractions were performed, each lasting ~3 s with 30 s rest between repetitions. The peak torque was determined as the maximal torque generated over the three repetitions. Participants were given visual feedback via the dynamometer monitor to maximise effort.

Muscle Soreness Muscle soreness was assessed via the use of a 200 mm visual analogue (VAS) and pain pressure threshold) PPT using a handheld pain algometer (Pain Test FPIX 50 Force One, Wagner Instruments, Greenwich, CT, USA) during visits 2-9. Participants rated their elbow flexor soreness during active flexion and extension of the elbow on the VAS; the far-left end point representing 'no pain' (0 mm) and the far-right end point representing 'unbearably painful' (200 mm). For PPT measures, participants were seated upright, with their arm rested at 90 degrees from full flexion. Application of increasing pressure of the algometer was applied via the probe through a 1 cm diameter head to the belly of the muscle , until the participants indicated the pain to be intolerable. At this point the force value (N) was recorded. Two measures were taken (2 cm apart ) at each site by the same investigator at baseline, 24, 48, and 72 h after completion of the damage protocol. The location of the measures were marked after the initial visit with a semi-permanent pen, in order to ensure consistency on the consecutive days. The mean of the two measures was used for data analysis (N).

Limb Girth An anthropometric tape measure (SciChem, Aberdeen, UK) was used to determine bicep circumference, whilst the arm was relaxed down by the participant's side. Mid-bicep circumference was determined by locating the mid-way between the acromion process and lateral epicondyle of the humerus. The mid-point was marked with a semi-permanent pen to ensure consistency on subsequent days. The same investigator took the average of two measurements; the technical error of measurement (TEM) was 0.29 cm (0.41 %).

Range of Motion (ROM) Joint ROM was determined by participants standing upright with their arm flexed at the shoulder and elbow. From this position, participants were asked to fully extend the limb until they were unable to move further without experiencing discomfort. The elbow joint angle was determined by using a goniometer and universal landmarks (the styloid process of the radius, lateral epicondyle of the humerus and the acromion process) to ensure correct alignment. The landmarks were marked with semi-permanent pen, so the goniometer could be placed in the same way on consecutive days. The same investigator took the average of two measurements; the TEM was 1.41 °(0.42 %).

Blood Sampling Procedure Venous blood samples were collected from the antecubital fossa at baseline, 24, 48 and 72 h post the damage protocol, before all other variables were assessed. Samples were immediately centrifuged (3000 × g) at 4°C for 15 min and the supernatant was aspirated into aliquots and then stored at -80 °C until analysis. Serum CK was analysed using an automated device (Cobas c702, Roche Diagnostics, Switzerland), with repeatability coefficient of variation 0.5 %.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Active

Exclusion Criteria:

* Food allergy
* Smokers
* Cardiovascular/gastrointestinal/thyroid/renal disease
* Musculoskeletal injury

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Maximal Voluntary Contraction | Measurements were taken on 8 separate occasions. Once at baseline, 24 hour 48 hours and 72 hours after the damage protocol (Bout 1) then repeated again for Bout 2, two weeks later.
  Maximal voluntary contraction measures the force capacity of the forearm flexor muscles

SECONDARY OUTCOMES:
Active Muscle Soreness | Measurements were taken on 8 separate occasions. Once at baseline, 24 hour 48 hours and 72 hours after the damage protocol (Bout 1) then repeated again for Bout 2, two weeks later.
  Visual analog scale to assess perceptual soreness, on a standard 200 mm line with the far-left end point representing 'no pain' (0 mm) and the far-right end point representing 'extremely painful' (200 mm).
Pain Pressure Threshold | Measurements were taken on 8 separate occasions. Once at baseline, 24 hour 48 hours and 72 hours after the damage protocol (Bout 1) then repeated again for Bout 2, two weeks later.
  For PPT measures, participants were seated upright, with their arm rested at 90 degrees from full flexion. Application of increasing pressure of the algometer was applied via the probe through a 1 cm diameter head to the belly of the muscle , until the participants indicated the pain to be intolerable. At this point the force value (N) was recorded.
Limb Girth | Measurements were taken on 8 separate occasions. Once at baseline, 24 hour 48 hours and 72 hours after the damage protocol (Bout 1) then repeated again for Bout 2, two weeks later.
  The girth of participants biceps were assessed to measure localised swelling with a tape measure.
Range of Motion | Measurements were taken on 8 separate occasions. Once at baseline, 24 hours 48 hours and 72 hours after the damage protocol (Bout 1) then repeated again for Bout 2, two weeks later.
  The range of motion participants could perform around their elbow joint was assessed to indirectly measure muscle damage, using a goniometer .
Serum Concentration of Creatine Kinase | Measurements were taken on 8 separate occasions. Once at baseline, 24 hours 48 hours and 72 hours after the damage protocol (Bout 1) then repeated again for Bout 2, two weeks later.
  Blood sample to measure indirect muscle damage

CONTACTS AND LOCATIONS:
Overall Officials: Glyn Howatson, Principal Investigator — Northumbria Univeristy
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No